CLINICAL TRIAL: NCT02074722
Title: Brain-Computer Interface and Mind-Body Awareness Training
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1312M46727
Record Dates: First submitted 2014-02-07; First posted 2014-02-28 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Subjects: Healthy Subjects

SUMMARY:
Mind-Body Awareness Training (MBAT), in the forms of various yoga and meditative practices, has become increasingly prevalent due to an increase in awareness of the potential health benefits, and improvements in concentration that this training can provide to practitioners. In the present study, we investigate the role of Mind-Body Awareness Training (MBAT) in the initial learning of a sensorimotor (SMR) based Brain-Computer Interface (BCI).

The PI's hypothesis is that MBAT will improve performance in SMR based BCI.

DETAILED DESCRIPTION:
In this protocol, we will test the PI's hypothesis that MBAT including yoga will improve the ability for subjects to concentrate on control the SMR thus improving the performance of BCI.

Subjects will be recruited for short term MBAT and then undergo BCI training. The performance of subjects with MBAT will be compared with those without MBAT to test the hypothesis. Procedures involved include 6 weeks yoga classes with at least 3 classes per week, and a EEG brain noninvasive brain computer interface study.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years old healthy subjects

Exclusion Criteria:

* History of traumatic brain injury/brain lesion, history of neurological deficit or neurodegenerative disorder, or history of epileptic seizures.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy population in Minneapolis area
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2014-03; Primary Completion 2017-06-28 (Actual); Study Completion 2017-06-28 (Actual)

PRIMARY OUTCOMES:
Performance over BCI sessions | one to three months
  During the course of the study over 5-10 weeks, we will quantitatively examine three main components of data: the proportion of subjects that achieve a pre-determined threshold of one-dimensional BCI competency as a time to event analysis, how subjects performed on average in each metric (accuracy, speed, etc.) over the course of the study (5-10 weeks), and subject learning over time during the course of study (5-10 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Bin He, PhD, Principal Investigator — University of Minnesota
Locations (1):
- Nils Hasselmo Hall at the University of Minnesota - Twin Cities Campus, Minneapolis, Minnesota, United States